CLINICAL TRIAL: NCT04757493
Title: The Effects of Prucalopride in Patients With Constipation Predominant Irritable Bowel Syndrome: A Double Blind Placebo Controlled Trial
Brief Title: The Effects of Prucalopride in Patients With Constipation Predominant Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Ovizit Saha, MD Resident, Gastroenterology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSMMU/2021/394
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — prucalopride

STUDY DESIGN:
Intervention Model Description: Its a randomized placebo controlled parallel group clinical trial. Prucalopride group is designated as "A" and placebo group is designated as group "B".
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant, care provider and primary outcome assessor will unaware about the allocated treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prucalopride group (A) (Active Comparator): Prucalopride 2 mg tablet, once daily in morning before breakfast will use as intervention in arm "A".
  Interventions: Drug: Prucalopride 2mg
- Placebo group (B) (Placebo Comparator): Placebo will be given at the same time and same dose in arm "B" . Both active drug and placebo have packed in the same type of strip.
  Interventions: Drug: Prucalopride 2mg

INTERVENTIONS:
Drug: Prucalopride 2mg — Both prucalopride 2mg and placebo will be administered for 6 weeks. Primary outcome will measure at 2nd and 6th week of treatment.
  Other Names: Placebo

SUMMARY:
Irritable bowel syndrome (IBS) is very common functional gastrointestinal disorder in daily gastrointestinal practice. Its etiology is multifactorial and incompletely understood. Different types of treatment have been trying but no single drug is effective for every patients. After the discovery of 5HT4(5 hydroxytryptamine-4) receptor and its effect on gastrointestinal motility, 5HT4 receptor agonist becoming a good therapeutic tool in different functional gastrointestinal disorder. Prucalopride is a selective 5HT4 agonist and it has proven benefit in chronic idiopathic constipation but there is not enough evidence that it is effective in constipation predominant IBS.

Objective: To assess the efficacy of Prucalopride in constipation predominant IBS patients.

Material & method: Consecutive patients of both sexes, age more than 18 years attended the outpatient department of Gastroenterology meeting the inclusion Criteria of IBS-C will be initially enrolled for the study. Their clinical history, examination & initial investigations report will be noted on the standard data sheet. Any alternative diagnosis if proven by clinical examination or laboratory investigation will be excluded from the study. Randomization into two groups (Prucalopride and placebo) will be performed by lottery. Patients will be randomly assigned to receive either Prucalopride 2 mg or placebo for 6 weeks. IBS symptoms will be assessed by IBS-SSS (symptom severity score) and IBS-QOL(quality of life) at the baseline, 2nd week and 6th week of treatment (end of treatment). Any adverse effect due to drugs will also be monitored by base line ECG, calculation of corrected QT interval and ECG monitoring (2 weeks and 6 weeks) during the course of treatment.

Data analysis By SPSS. IBS-SSS and IBS-QOL instrument scores will be expressed as mean ± standard deviation. Statistical analysis will be done by paired and unpaired 't' test. P value <0.05 will be considered statistically significant.

Ethical Consideration:

Every ethical issue will be discussed with the patient regarding the study and informed written consent will be obtained. There will be no chance of disclosure of information that will have been harmful to the patients or others. Permission have been taken from the concerned departmental ethical committee as well as ethical review committee of BSMMU in order to carry out the study.

DETAILED DESCRIPTION:
Consecutive patients of both sexes, age more than 18 years attended the outpatient department of Gastroenterology meeting the inclusion Criteria of IBS-C will be initially enrolled for the study. Their clinical history, examination & initial investigations with Complete Blood Count , C-Reactive Protein, Tissue Transglutaminase antibody, Oral Glucose Tolerance Test, Thyroid Stimulating Hormone will be done from respected department of BSMMU. Report will be noted in the standard data sheet. Any alternative diagnosis if proven by clinical examination or laboratory investigation will be excluded from the study. All participants will be advised to maintain their usual dietary practices throughout the study. The subject will be recruited according to sample size. Total study population will be divided in to Prucalopride and placebo group. An independent treatment code will be generated and allocated according to sample size in each group. Randomization into two groups will be performed by lottery. The independent treatment codes and allocation will be maintained, which will be locked until all analyses will have been completed. Thus, the clinical trial will be performed double-blind with all patients and investigators will unaware of which treatment is allocated.

One group will receive tab Prucalopride 2 mg once daily 30 minute before breakfast, while the other group will receive identical looking placebo one tab once daily at same time. The tablets will be administered for a total of 6 weeks. Before starting treatment each individual will undergo a baseline assessment during which demographic data, base line investigations, IBS symptoms by IBS-SSS and QOL data will be recorded. Patients will be followed-up at 2 weeks, then at 6 weeks by IBS-SSS questionnaire and IBS-QOL questionnaire. Patients will be asked to return with the strips of the ingested drugs at the end of the treatment to count & ensure compliance. Any adverse effect due to drugs will also be monitored by base line ECG, calculation of corrected QT interval and ECG monitoring (2 weeks and 6 weeks) during the course of treatment. Any adverse event will be responded quickly and documented at the same time.

IBS-SSS is a 5 item tools. It is primarily a measure of IBS symptoms including abdominal pain and distension as well as bowel satisfaction. This scale evaluates IBS symptoms: abdominal pain, abdominal distension, stool frequency and consistency and interference with life in general. The IBS-SSS calculates the sum of these 5 items scored on a visual analogue scale from 0-100. Determination of severity of each symptom is determined by the patient. The nature of the items on IBS-SSS is appropriate to be used in clinical trials. The items are summed and thus the total score can range from 0 to 500 points. IBS severity has the following defined ranges: mild 75-174, moderate 175-300, and severe > 300.

The IBS-QOL questionnaire is a 34-item instruments which assess QOL impairment due to IBS symptoms. Each item is scored on a five-point scale (1 = not at all, 5 = extremely) that represents one of eight dimensions (dysphoria, interference with activity, body image, health-related worries, food avoidance, social reactions, sexual dysfunction, and relationships). After scoring by the patient, responses will be transformed to reverse code system (5= not at all, 1= extremely). Items are scored to derive an overall total score of IBS related QOL. To facilitate score interpretation, the summed total score is transformed to a 0-100 scale ranging from zero (poor QOL) to 100 (maximum QOL). The QOL instrument will be given to each patient before treatment is started. The patient will complete the form according to schedule and all data will be recorded and entered onto a data sheet.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-65 years.
* Patients who will Meet Rome IV criteria for IBS-Constipation (IBS-C).
* Patients classified as IBS-C had > 25% hard or lumpy stool (Bristol stool scale 1-2) and < 25% loose or watery (Bristol stool scale 6-7).
* Absence of alarm features (rectal bleeding, anemia, unexplained weight loss, and a family history of organic GI diseases (e.g. colon cancer or inflammatory bowel disease).
* Patients more than 55 years when full colonoscopy will normal.
* Patients given informed written consent.

Exclusion Criteria:

* Current treatment with laxative and Selective Serotonin Re-uptake Inhibitor.
* Unable or Unwilling to stop medication including lactulose, lubiprostone etc.
* Known organic bowel diseases (e.g. inflammatory bowel disease, tuberculosis, diverticular disease, etc.).
* Secondary causes of constipation e.g. Diabetes Mellitus, Hypothyroidism, Cerebrovascular disease and Parkinsonism. Known severe depression and psychiatric disorder.
* Clinical feature suggestive of organic disease (H/O weight loss, per rectal bleeding, family history of malignancy etc).
* Previous GI surgery.
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Assess the Change of IBS symptoms from baseline by using IBS-Symptom Severity Score | Base line, during treatment (2nd week) and after 6 weeks
  IBS-Symptom Severity Score is a 5 item tools.This scale evaluates IBS symptoms: abdominal pain, abdominal distension, stool frequency and consistency and interference with life in general. The IBS-Symptom Severity Score calculates the sum of these 5 items scored on a visual analogue scale from 0-100. Determination of severity of each symptom is determined by the patient.The items are summed and thus the total score can range from 0 to 500 points. IBS severity has the following defined ranges: mild 75-174, moderate 175-300, and severe > 300. Improvement is defined as decrease of 50 points from baseline.
Assess the change of quality of life from baseline by using IBS- Quality of life questionnaire | Base line, during treatment (2nd week) and after 6 weeks
  IBS-Quality of life instrument contains 34 question items relating to symptoms of IBS. The magnitude of the respondents feelings to each item is determined by the patients selection of the five Likert-style responses.Responses are transformed to reverse code system. The total score is transformed to 0-100 scale where 0 means poor quality of life and 100 means maximum quality of life. Ten(10) points improvement from base line will be considered clinically meaningful improvement

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr. Anwarul Kabir, MD, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Shahbag, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No